CLINICAL TRIAL: NCT03580174
Title: Investigation of the Effects of Physiotherapy and Rehabilitation Programs Following Botulinum Toxin Injection on Body Functions, Activity and Participation in Children With Cerebral Palsy
Brief Title: The Effects of Physiotherapy and Rehabilitation Programs Following Botulinum Toxin on Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Kübra Seyhan, Research Assisstant, MSc, PT, Hacettepe University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 57/30
Record Dates: First submitted 2018-05-31; First posted 2018-07-09 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Cerebral Palsy
Keywords: Physical therapy; ICF; Botulinum toxin; Activity; Function
MeSH Terms: conditions — Cerebral Palsy; Motor Activity

STUDY DESIGN:
Intervention Model Description: There will be two groups as Routine Physiotherapy group and Goal Directed Activity Based Physical Therapy (GDPT) group.
  * Routine Physiotherapy (RPT) group: Ten children with CP will RPT applications will consist of unstructured stretching exercises, massage, passive range of motions, muscle strengthening, orthotics etc.) .
  * Goal Directed Activity Based Physical Therapy (GDPT) group: Ten children with CP will receive structural, comprehensive activity based, goal directed therapy protocol one hour in a session, 2 times in a week during 8 weeks. GDPT will be a structural protocol and consists of daily life activities as sit to stand and reach, treadmill exercises, balance exercises with bosu-ball, orthotics, home program, following with exercise-diary.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Goal directed physiotherapy group (Active Comparator): Ten children with CP will receive structural, comprehensive activity based, goal directed physiotherapy
  Interventions: Other: Goal directed physiotherapy group
- Routine physiotherapy group (Active Comparator): Ten children with CP will receive conventional, traditional physiotherapy
  Interventions: Other: Routine physiotherapy group

INTERVENTIONS:
Other: Goal directed physiotherapy group — Ten children with CP will receive structural, comprehensive activity based, goal directed therapy protocol one hour in a session, 2 times in a week during 8 weeks. GDPT will be a structural protocol and consists of daily life activities as sit to stand and reach, treadmill exercises, balance exercises with bosu-ball, orthotics, home program, following with exercise-diary.
  Arms: Goal directed physiotherapy group
Other: Routine physiotherapy group — Ten children with CP will RPT applications will consist of unstructured stretching exercises, massage, passive range of motions, muscle strengthening, orthotics etc.) one hour in a session, 2 times in a week during 8 weeks.
  Arms: Routine physiotherapy group

SUMMARY:
The purpose of this study was to investigate the effects of Physiotherapy and rehabilitation program on body functions and structures, activity and participation levels, personal and environmental factors following Multilevel Botulinum toxin (BT) injections on ambulatory children with Cerebral Palsy (CP). Two physiotherapy and rehabilitation methods which are structural goal directed activity based physiotherapy (intervention group; 10 children with ambulatory Cerebral Palsy) and unstructured routine physiotherapy (control group; 10 children with ambulatory Cerebral Palsy) will be compared.

DETAILED DESCRIPTION:
The purpose of this study was to investigate the effects of Physiotherapy and rehabilitation program following Multilevel Botulinum toxin (BT) injections on ambulatory children with Cerebral Palsy (CP). Children who are 3-12 years, have Diplegic CP, able to walk with/without support (between GMFCS level I-III), have multilevel botulinum toxin injections to lower extremity muscles, able to communicate, whose parents agree to participate will include in this study. Children who had lower extremity surgery in last six months, who have repeated BT during the study, do not want to continue the study will exclude the current study. It is planned to receive at least 20 children with CP. Children will be divided into two groups: ten children in routine physiotherapy (RPT) group (traditional methods, stretch, massage etc.) and ten children in goal directed activity based physical therapy (GDPT) group (structural concept).

Routine Physiotherapy (RPT) group: Ten children with CP will RPT applications will consist of unstructured stretching exercises, massage, passive range of motions, muscle strengthening, orthotics etc.) .

Goal Directed Activity Based Physical Therapy (GDPT) group: Ten children with CP will receive structural, comprehensive activity based, goal directed therapy protocol one hour in a session, 2 times in a week during 8 weeks. GDPT will be a structural protocol and consists of daily life activities as sit to stand and reach, treadmill exercises, balance exercises with bosu-ball, orthotics, home program, following with exercise-diary.

Hypothesis 1: GDPT program applied after multilevel BT injection in children with CP affects the body structure and functions.

Hypothesis 2: GDPT program applied after multilevel BT injection in children with CP affects the activity.

Hypothesis 3: GDPT program applied after multilevel BT injection in children with CP affects the participation.

Hypothesis 4: GDPT after BT injection in children with CP affects the activity of the child more than RPT.

The first evaluation will be made in the first week after BT injection. After 8 weeks therapy program is applied, the second evaluation will be made.

The assessments to be implemented under the International Classification of Functioning (ICF) framework are as follows:

Body structure and functions

* Muscle tone (Modified Ashworth Scale-MAS)
* Muscle Strength (with Manual Muscle Tester Device)
* Lower Extremity Selective Motor Control (Selective Control Assessment of Lower Extremity- SCALE)
* Spatiotemporal characteristics of gait (Gait trainer)

Activity and participation:

* Balance (Pediatric Balance Scale- PBS)

  . Trunk Control (Trunk Control Measurement Scale -TCMS)
* Pediatric Evaluation of Disability Inventory (PEDI)
* Gait Analysis (Modified Physician Rating Scale (MPRS); Gillette Functional Gait Assessment)
* Motor Function (Gross Motor Function Measurement -GMFM)

Personal and Environmental Factors:

Level of anxiety and satisfaction of parents and children will be rated between 11-point scale on self reported questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* 3-12 years,
* have Diplegic CP
* able to walk with/without support (between GMFCS level I-III)
* have multilevel botulinum toxin injections to lower extremity muscles
* able to communicate
* whose parents agree to participate

Exclusion Criteria:

* who had lower extremity surgery in last six months
* who have repeated BT during the study
* do not want to continue the study

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-05-05 (Actual); Study Completion 2019-06-18 (Actual)

PRIMARY OUTCOMES:
Modified Physician Rating Scale | 10 minutes
  The Modified Physicians' Rating Scale (MPRS) is an observational tool that has been used to evaluate gait and assess the outcome of botulinum toxin injection in children with cerebral palsy. This is a scale adapted from the Physicians rating scale which was created to examine the gait of children with CP in the sagittal plane after botulinum toxin A for equinus gait. It is a scale with 8 sections where you score both the left and right lower extremity from video record of child's gait. The score ranged 0 to 22 point. A perfect score would be a 22 on each limb. MPRS should be observed from front and sides of children with CP.

SECONDARY OUTCOMES:
Manual Muscle Test | 10 min
  Manual muscle tester (hand held dynamometer) will use for quantifying objectively strength of lower extremity muscles. Dynamometry provides an objective measure of isometric strength against examiner resistance by quantifying the mechanical force or torque. Hand-held dynamometry (HHD) was used to measure the force (in Newtons) generated during an isometric contraction. This device records force for intervals of 0.1 N up to a maximum 99.9 N, thereafter in whole Newtons. These were recorded in order, as trials 1 to 3.
Gait Analysis | 10 min
  Spatiotemporal gait deviation of children will be evaluated with Biodex Gait Trainer 2 like as a treadmill gait analysis. The device will give us about "Average Walking Speed, Average Step Cycle, Average Step Length, Coefficient of Variance, Right/left time distribution, Ambulation Index. The composite score's goal is 100. The higher point is the better.
Gillette Functional Gait Assessment | 5 min
  Level of locomotion will assess with Gillette Functional Gait Assessment that was a 10-level, parent-report walking scale and encompassing a range of walking abilities from nonambulatory to ambulatory in all community settings and terrains was developed at Gillette Children's Specialty Healthcare (GCSH) as part of the Gillette Functional Assessment Questionnaire (FAQ). Gait was ranged between 1 to 10 level. The high point determined better locomotion level.
Pediatric Balance Scale | 5 min
  Balance will evaluated with Pediatric Balance Scale (PBS). It has 14 item. Maximum point 56 points with 56 points being a perfect score.
Gross Motor Function Measurement | 15 min
  Motor Functions of children will be evaluated with Gross Motor Function Measurement (GMFM). It is a clinical tool designed to evaluate change in gross motor function in children with cerebral palsy.There is 88 items under 5 subdimensions (lying and rolling, sitting, crawling and kneeling, standing, walking-running-jumping) with a 4-point scoring system for each item. The percentage of sub-dimensions and total scores calculated separately. The higher percentage score (ranged between 0-100 point) was the better gross motor function.
Parent-reported questionnaire | 2 min
  We prepare a questionnaire for asking the level of anxiety and satisfaction of parents. The 11-point numeric scale ranges from '0' representing parent feeling negatively to '10' representing parent feeling positively.
Modified Ashworth Scale | 5 min
  Tone of lower extremity muscles will be assessed with Modified Ashworth Scale. The Modified Ashworth scale s (MAS) is the most frequently cited of the available clinical rating scales to measure tonal abnormality. It is already being used to evaluate the effects of drug treatments for spasticity. The spasticity of each muscle ranged between 0 to 5. (0:No increase in muscle tone,1:Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is(are) moved in flexion or extension, 2: Slight increase in muscle tone, manifested by a catch followed by minimal resistance through the remainder of the range of motion but the affected part(s) is(are) easily moved, 3;More marked increase in muscle tone through most of the range of movement, but affected part(s) easily moved, 4:Considerable increase in muscle tone, passive movement difficult, 5:Affected part(s) is(are) rigid in flexion or extension).
Selective Control Assessment of Lower Extremity | 3 min
  Lower Extremity Selective Motor Control will be evaluated with Selective Control Assessment of Lower Extremity (SCALE). The SCALE tool was designed for clinical administration and scoring by health car e professionals, to be used without specialized equipment. The tool includes 'Directions for Administration,' 'Instructions for Grading,' and a 'Score Sheet.' Hip , knee, ankle, sub-talar, and toe joints are assessed bilaterally. Selective movement control is graded at each joint as 'Normal' (2 points), 'Impaired' (1 point), or 'Unable' (0 points). The higher point is the better selectivity of movement.
Trunk Control Measurement Scale | 15 min
  Trunk Control will be assessed with Trunk Control Measurement Scale (TCMS) in children with CP. The TCMS divided three sub-dimensions like as static sitting balance, selective movement control and dynamic reaching. The maximum value for the total TCMS is 58 (20 points for the category static sitting balance, 28 points for selective movement control and 10 for dynamic reaching). A higher TCMS scores indicates a better performance in trunk control.

CONTACTS AND LOCATIONS:
Overall Officials: Mintaze GÜNEL, Prof., Study Director — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Sıhhıye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Biyik KS, Gunel MK, Akyuz EU. How does treadmill training contribute to botulinum toxin application plus routine physical therapy in ambulatory children with spastic bilateral cerebral palsy? A randomized controlled trial. Ir J Med Sci. 2023 Feb;192(1):209-217. doi: 10.1007/s11845-022-02960-9. Epub 2022 Feb 27. PMID 35224682